CLINICAL TRIAL: NCT00000613
Title: CVD Risk and Health in Postmenopausal Phytoestrogen Users
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 116; R01HL057790 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2005-12

CONDITIONS: Bone Diseases; Cardiovascular Diseases; Coronary Disease; Depression; Heart Diseases; Myocardial Ischemia; Osteoporosis; Postmenopause
MeSH Terms: conditions — Bone Diseases; Cardiovascular Diseases; Coronary Disease; Depression; Heart Diseases; Myocardial Ischemia; Osteoporosis | interventions — Dietary Supplements; Genistein; Diet; Soybean Proteins

INTERVENTIONS:
Behavioral: dietary supplements
Drug: genistein
Behavioral: diet, soy proteins

SUMMARY:
To determine the acceptability and benefits of use of a dietary supplement of the phytoestrogen, genistein, versus placebo on heart disease risk factors, bone density, and psychosocial outcomes in postmenopausal women.

DETAILED DESCRIPTION:
BACKGROUND:

Estrogen replacement therapy is beneficial for heart disease risk factors as well as for bone density. However, a large proportion of postmenopausal women are not compliant with therapeutic regimens. Phytoestrogens are naturally occurring compounds found in plants and soy products that have estrogenic effects, and may represent an alternative treatment for the prevention of heart disease and osteoporosis in postmenopausal women. However, few intervention trials have examined the extent to which it is possible to improve heart disease risk factors, bone density, and quality of life in postmenopausal women through use of a dietary supplement of phytoestrogen.

DESIGN NARRATIVE:

Randomized, double-blind, placebo-controlled study. A total of 210 women were enrolled in the study to be followed for one to two years. The women were randomized to phytoestrogen treatment or to placebo. Data are collected at baseline visits, at one and three month follow-up telephone calls, and at 6, 12, and 24 month follow-up clinic visits. Measures of high density lipoprotein and other heart disease risk factors, hip and spine bone density, and depression, life satisfaction, and quality of well-being are obtained. Cross-sectional and longitudinal comparisons of treatment and placebo groups are performed before and after adjustment and stratification for potentially confounding covariates.

The study was renewed in March 2002 to assess whether the women treated with phytoestrogens had lowered homocysteine, interleukin-6, C-reactive protein, E-selectin, and decreased obesity and fat mass over two years.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Postmenopausal women, ages 45 to 74.

Ages: 45 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-04; Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Kritz-Silverstein — University of California, San Diego

REFERENCES:
- [Background] Goodman-Gruen D, Kritz-Silverstein D. Usual dietary isoflavone intake is associated with cardiovascular disease risk factors in postmenopausal women. J Nutr. 2001 Apr;131(4):1202-6. doi: 10.1093/jn/131.4.1202. PMID 11285326
- [Background] Kritz-Silverstein D, Goodman-Gruen DL. Usual dietary isoflavone intake, bone mineral density, and bone metabolism in postmenopausal women. J Womens Health Gend Based Med. 2002 Jan-Feb;11(1):69-78. doi: 10.1089/152460902753473480. PMID 11860727
- [Background] Goodman-Gruen D, Kritz-Silverstein D. Usual dietary isoflavone intake and body composition in postmenopausal women. Menopause. 2003 Sep-Oct;10(5):427-32. doi: 10.1097/01.GME.0000058866.35869.B4. PMID 14501604